CLINICAL TRIAL: NCT06944912
Title: Combined Transversalis Fascia and Transversus Abdominis Plane Blocks Versus Intrathecal Morphine: Effects on Postoperative Opioid Consumption and Obstetric Recovery After Cesarean Section
Brief Title: Transversus Abdominis and Transversalis Fascia Plane Block Combination for Cesarean Section
Acronym: TAPTFPB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ali Ahiskalioglu, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUTFTAPTFP
Record Dates: First submitted 2025-04-18; First posted 2025-04-25 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Ceserean Section and Postoperative Pain
Keywords: Postoperative Recovery; Cesarean Section; Postoperative Pain; Transversalis Fascia Plane Block; Transversus Abdominis Plane Block; Intrathecal Opioid; ObsQoR-10 T
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transversalis fascia+Transversus abominis plane block (Active Comparator)
  Interventions: Procedure: Transversalis fascia plane block and transversus abdominis plane block
- Intrathecal Morphine (Active Comparator)
  Interventions: Procedure: Intrathecal Morphine

INTERVENTIONS:
Procedure: Transversalis fascia plane block and transversus abdominis plane block — 20 ml local anesthetics for Transversus Abdominis Plane block and 10 ml local anesthetics for Trasnversalis fascia plane block
  Arms: Transversalis fascia+Transversus abominis plane block
Procedure: Intrathecal Morphine — 100 mcg morphine with local anesthetics injected intrathecally
  Arms: Intrathecal Morphine

SUMMARY:
Cesarean delivery rates are rising globally, and effective postoperative analgesia is crucial for maternal recovery and newborn care. While intrathecal morphine offers strong analgesia, it may cause side effects such as nausea, pruritus, or respiratory depression. The transversus abdominis plane (TAP) block provides somatic pain relief but is often insufficient alone. The transversalis fascia plane block (TFPB) has been shown to enhance lower abdominal analgesia. This study aims to evaluate whether combining TAP and TFP blocks can provide analgesic efficacy comparable to intrathecal morphine in cesarean section patients who are unable to receive opioids or are at high risk of side effects.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* American Society of Anesthesiologists physical score I or II
* caesarean section with a Pfannenstiel incision

Exclusion Criteria:

* additional surgical intervention, or received general anaesthesia,
* hypersensitivity to the agents to be used
* BMI greater than 35 kg m-2
* coagulopathy,
* local infection,
* opioid addiction,
* pregnancy-related hypertension
* diabetes mellitus

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
The Obstetric Quality of Recovery-10 (ObsQoR-10) Score | Postoperative 24 hours
  The questionnaire's subscales are physical comfort (n=3 items), emotional state (n=2 items), pain (n=1 item), physical independence (n=2 items), and the ability to take care of the newborn (n=2 items). Each item is scored on a scale of 0-10, except for the first four items, which are graduated from 10 to 0. The total score is the sum of all item scores (i.e. a score ranging from 0 to 100, where 0 is the worst recovery score, and 100 indicates the best).

SECONDARY OUTCOMES:
Opioid consumption | Postoperative 24. hours
  Patient controlled analgesia based opioid requirement

CONTACTS AND LOCATIONS:
Overall Officials: Ali Ahiskalioglu, Prof., Principal Investigator — Atatürk University, Faculty of Medicine, Department of Anesthesiology and Reanimation
Locations (1):
- Atatürk University Hospital, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pinarbasi A, Altiparmak B, Korkmaz Toker M, Pirincci F, Ugur B. Ultrasound-guided transversalis fascia plane block or transversus abdominis plane block for recovery after caesarean section: A randomised clinical trial. Eur J Anaesthesiol. 2024 Oct 1;41(10):769-778. doi: 10.1097/EJA.0000000000002041. Epub 2024 Jul 22. PMID 39039833
- [Result] Aydin ME, Bedir Z, Yayik AM, Celik EC, Ates I, Ahiskalioglu EO, Ahiskalioglu A. Subarachnoid block and ultrasound-guided transversalis fascia plane block for caesarean section: A randomised, double-blind, placebo-controlled trial. Eur J Anaesthesiol. 2020 Sep;37(9):765-772. doi: 10.1097/EJA.0000000000001222. PMID 32412986
- [Derived] Cadirci DY, Aydin ME, Ahiskalioglu EO, Celik EC, Yayik AM, Coruh S, Senocak GNC, Ciftci B, Ahiskalioglu A. Intrathecal morphine versus transversalis fascia and transversus abdominis plane blocks combination on obstetric quality of recovery after cesarean delivery: a randomized controlled trial. BMC Anesthesiol. 2025 Dec 17. doi: 10.1186/s12871-025-03559-0. Online ahead of print. PMID 41408168